CLINICAL TRIAL: NCT06450600
Title: Enhancing Quality of Life in Multiple Sclerosis: a Study Protocol to Evaluate the Impact of a Therapeutic Education Program
Brief Title: Enhancing Quality of Life in MS Patients Through Tailored Therapeutic Education
Acronym: MS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Akhrif Iman (Other Government)
Responsible Party: Sponsor-Investigator, Akhrif Iman, Principal Investigator, Ibn Sina Hospital
Organization: Ibn Sina Hospital (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: u7f528ek
Record Dates: First submitted 2024-04-03; First posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-04

CONDITIONS: Multiple Sclerosis (MS)
Keywords: Multiple Sclerosis; therapeutic education program; bladder dysfunction
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: This study is an observational, descriptive, and analytical research without a control group, aimed at assessing the impact of a specialized therapeutic education program on the quality of life of patients with multiple sclerosis. Participants will receive individual sessions to assess their needs, followed by targeted educational workshops on various aspects of disease management. The effectiveness of the program will be primarily measured using the Multiple Sclerosis Quality of Life-54 (MSQOL-54) questionnaire, with secondary outcomes assessed by the Urinary Handicap Measure (M.H.U) scale.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Therapeutic Education Program for Multiple Sclerosis Patients (Experimental): Participants in this arm will receive a comprehensive therapeutic education program designed specifically for individuals diagnosed with multiple sclerosis. The program includes individual assessments to identify patient needs and concerns, followed by targeted educational workshops. These workshops cover a wide range of topics, including disease understanding, bladder and sphincter management, fatigue management, and psychological well-being. The intervention is delivered by a multidisciplinary team, including physiotherapists, neurologists, psychologists, urologists, occupational therapists, nurses, and nutritionists, aiming to improve participants' quality of life by enhancing their disease management skills and overall well-being.
  Interventions: Behavioral: Multiple Sclerosis Therapeutic Education Program

INTERVENTIONS:
Behavioral: Multiple Sclerosis Therapeutic Education Program — The "MS Self-Management Education Workshop" is designed as an integral part of our therapeutic education program targeting individuals diagnosed with multiple sclerosis (MS). This intervention focuses on empowering participants with knowledge and skills necessary for effective self-management of their condition. The workshop includes interactive sessions that cover a range of topics critical for MS patients, such as:
  Understanding the nature and progression of MS, highlighting the importance of early symptom recognition and management strategies.
  Techniques for managing common MS symptoms, including fatigue, mobility issues, and cognitive challenges, with practical advice on daily living adaptations.
  Guidance on medication management, including the use of disease-modifying therapies and managing side effects.
  Strategies for emotional well-being, including coping mechanisms for dealing with the psychological impact of MS, stress management, and fostering resilience.
  Other Names: MS Self-Management Education Workshop

SUMMARY:
Within the framework of improving the quality of life for patients with Multiple Sclerosis (MS), this prospective and descriptive study aims to evaluate the effectiveness of a therapeutic education program. The program, designed specifically for MS patients, includes individual sessions to identify needs, fears, and questions, followed by targeted educational workshops. These workshops address understanding the disease, managing bladder and sphincter issues, fatigue management, and psychological well-being, relying on a multidisciplinary team including physiotherapists, neurologists, psychologists, urologists, occupational therapists, nurses, and nutritionists. The primary goal is to assess the impact of this program on the quality of life of patients, measured by the MSQOL-54 questionnaire, with secondary measures such as the Urinary Handicap Scale (M.H.U). Fifty patients will be recruited from the Department of Physical Medicine and Rehabilitation at Rabat University Hospital, Morocco, with follow-ups planned at 3 and 6 months. This program aims to provide patients with the knowledge and skills necessary for better management of their condition, thereby promoting active participation in treatment and a significant improvement in their quality of life.

DETAILED DESCRIPTION:
This is a prospective, descriptive, and analytical study without a control group, aiming to measure the impact of a specialized therapeutic education program on the quality of life in individuals diagnosed with multiple sclerosis.

The educational program includes individual sessions to assess patient needs, followed by workshops facilitated by a multidisciplinary team. These workshops are designed to provide comprehensive support and education on various aspects of living with multiple sclerosis.

Understanding the Disease: This workshop will provide participants with a detailed understanding of multiple sclerosis, including its etiology, pathophysiology, and common symptoms. Participants will learn about the importance of early diagnosis, disease progression, and treatment options available.

Managing Bladder and Sphincter Issues: Bladder and sphincter dysfunction are common symptoms of multiple sclerosis that significantly impact quality of life. This workshop will focus on strategies for managing urinary symptoms, including bladder retraining, pelvic floor exercises, and the use of assistive devices. Participants will also receive guidance on managing bowel dysfunction and preventing complications such as urinary tract infections.

Fatigue Management: Fatigue is a pervasive and debilitating symptom of multiple sclerosis. This workshop will explore the causes of fatigue in MS and provide practical strategies for conserving energy and managing daily activities. Participants will learn about pacing techniques, energy-saving devices, and the importance of restorative sleep.

Psychological Well-being: Living with multiple sclerosis can have a significant impact on mental health and emotional well-being. This workshop will address coping strategies for managing stress, anxiety, and depression associated with the disease. Participants will learn relaxation techniques, mindfulness exercises, and how to access support services and community resources.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older Patients diagnosed with confirmed multiple sclerosis by a neurologist

Exclusion Criteria:

* Cognitive disorders Refusal to participate Significant visual impairments

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-05 (Estimated); Primary Completion 2025-04-05 (Estimated); Study Completion 2025-06-05 (Estimated)

PRIMARY OUTCOMES:
Multiple Sclerosis Quality of Life-54 (MSQOL-54) | The MSQOL-54 will be administered at the time of inclusion, 3 months after the initiation of the therapeutic education program, and again at 6 months after the initiation of the program.
  The MSQOL-54 is a multidimensional questionnaire specifically designed to assess the health-related quality of life of patients with multiple sclerosis. It comprises 54 items, each rated from 0 to 100, grouped into 12 dimensions with two independent questions. These dimensions include physical activity, limitations due to physical health, limitations due to emotional state, pain, emotional well-being, energy, perceived health, social function, cognitive function, distress, sexual function, and general well-being.

SECONDARY OUTCOMES:
Measure of Urinary Handicap scale (M.H.U) | The M.H.U will be administered at the time of inclusion, 3 months after the initiation of the therapeutic education program, and again at 6 months after the initiation of the program.
  The Measure of Urinary Handicap scale (M.H.U) is an assessment tool designed to measure the impact of urinary symptoms on individuals' quality of life. It typically consists of several questions that explore the frequency, severity, and psychosocial impact of urinary symptoms on a person's daily life. The responses to these questions allow for the generation of a score that reflects the degree of handicap or discomfort experienced by the patient due to their urinary symptoms.

IPD SHARING:
Plan to Share IPD: Yes
Study Objective: Develop and evaluate a structured educational program for MS patients to enhance quality of life. Design: Prospective study assessing program impact without a control group. Recruitment: From Rabat University Hospital's PRM and Neurology sessions. Intervention: Individual needs assessment followed by multidisciplinary-led educational workshops. Assessment: Patients evaluated at baseline, 3 and 6 months using MSQOL-54 and M.H.U scale. Outcome Measures: Primary: MSQOL-54 for quality of life. Secondary: M.H.U scale for urinary symptoms. Sample Size: Fifty patients recruited, considering 10% follow-up loss rate. Follow-up: Patients can withdraw at any time. Statistical Analysis: Collaboration with Epidemiology and Clinical Research Laboratory.
Supporting Information: Study Protocol
Time Frame: Day 0 (Baseline Assessment):
  Month 3 (3-Month Follow-up)
  Month 6 (6-Month Follow-up):
Access Criteria: Inclusion: Age 18+, confirmed MS diagnosis, ability to provide consent, and available for program and assessments. Exclusion: Cognitive impairment, refusal, significant visual impairment.

REFERENCES:
- [Background] Lotfi R, El Kardoudi A, Chigr F. Multiple sclerosis in Morocco: Epidemiological, clinical, and therapeutic profile. Mult Scler Relat Disord. 2024 Jan;81:105347. doi: 10.1016/j.msard.2023.105347. Epub 2023 Dec 2. PMID 38061315
- [Background] Ouadghiri S, El Alaoui Toussi K, Brick C, Ait Benhaddou EH, Benseffaj N, Benomar A, El Yahyaoui M, Essakalli M. Genetic factors and multiple sclerosis in the Moroccan population: a role for HLA class II. Pathol Biol (Paris). 2013 Dec;61(6):259-63. doi: 10.1016/j.patbio.2013.05.002. Epub 2013 Jul 9. PMID 23849771
- [Background] Dobson R, Giovannoni G. Multiple sclerosis - a review. Eur J Neurol. 2019 Jan;26(1):27-40. doi: 10.1111/ene.13819. Epub 2018 Nov 18. PMID 30300457
- [Background] McGinley MP, Goldschmidt CH, Rae-Grant AD. Diagnosis and Treatment of Multiple Sclerosis: A Review. JAMA. 2021 Feb 23;325(8):765-779. doi: 10.1001/jama.2020.26858. PMID 33620411
- [Background] El Alaoui Taoussi K, Ait Ben Haddou E, Benomar A, Abouqal R, Yahyaoui M. [Quality of life and multiple sclerosis: Arabic language translation and transcultural adaptation of "MSQOL-54"]. Rev Neurol (Paris). 2012 May;168(5):444-9. doi: 10.1016/j.neurol.2011.10.011. Epub 2012 May 2. French. PMID 22560010
- [Background] Palacios S, Ramirez M, Lilue M, Vega B. Evaluation of Femaxeen(R) for control of urinary incontinence in women: A randomized, double-blind, placebo-controlled study. Maturitas. 2020 Mar;133:1-6. doi: 10.1016/j.maturitas.2019.12.008. Epub 2019 Dec 16. PMID 32005419
- [Background] Demaille-Wlodyka S, Donze C, Givron P, Gallien P; ETP Sofmer Group. Self care programs and multiple sclerosis: physical therapeutics treatment - literature review. Ann Phys Rehabil Med. 2011 Mar;54(2):109-28. doi: 10.1016/j.rehab.2011.01.003. Epub 2011 Feb 18. English, French. PMID 21388907
- [Background] Perneger TV, Sudre P, Muntner P, Uldry C, Courteheuse C, Naef AF, Jacquemet S, Nicod L, Rochat T, Assal JP. Effect of patient education on self-management skills and health status in patients with asthma: a randomized trial. Am J Med. 2002 Jul;113(1):7-14. doi: 10.1016/s0002-9343(02)01136-1. PMID 12106617
- [Background] Stuifbergen AK. Health-promoting behaviors and quality of life among individuals with multiple sclerosis. Sch Inq Nurs Pract. 1995 Spring;9(1):31-50; discussion 51-5. PMID 7777743
- [Background] Acquadro C, Lafortune L, Mear I. Quality of life in multiple sclerosis: translation in French Canadian of the MSQoL-54. Health Qual Life Outcomes. 2003 Nov 24;1:70. doi: 10.1186/1477-7525-1-70. PMID 14636427
- [Background] Giordano A, Testa S, Bassi M, Cilia S, Bertolotto A, Quartuccio ME, Pietrolongo E, Falautano M, Grobberio M, Niccolai C, Allegri B, Viterbo RG, Confalonieri P, Giovannetti AM, Cocco E, Grasso MG, Lugaresi A, Ferriani E, Nocentini U, Zaffaroni M, De Livera A, Jelinek G, Solari A, Rosato R. Viability of a MSQOL-54 general health-related quality of life score using bifactor model. Health Qual Life Outcomes. 2021 Sep 25;19(1):224. doi: 10.1186/s12955-021-01857-y. PMID 34563229
- [Background] Stern B, Hojs Fabjan T, Rener-Sitar K, Zaletel-Kragelj L. Validation of The Slovenian Version of Multiple Sclerosis Quality of Life (MSQOL-54) Instrument. Zdr Varst. 2017 Oct 9;56(4):260-267. doi: 10.1515/sjph-2017-0035. eCollection 2017 Oct. PMID 29062401
- [Background] Rotstein D, Montalban X. Reaching an evidence-based prognosis for personalized treatment of multiple sclerosis. Nat Rev Neurol. 2019 May;15(5):287-300. doi: 10.1038/s41582-019-0170-8. PMID 30940920
- [Background] Kaya T, Goksel Karatepe A, Atici Ozturk P, Gunaydin R. Impact of peer-led group education on the quality of life in patients with ankylosing spondylitis. Int J Rheum Dis. 2016 Feb;19(2):184-91. doi: 10.1111/1756-185X.12256. Epub 2013 Dec 14. PMID 24330320
- [Background] Song Y, Xie X, Chen Y, Wang Y, Yang H, Nie A, Chen H. The effects of WeChat-based educational intervention in patients with ankylosing spondylitis: a randomized controlled trail. Arthritis Res Ther. 2021 Mar 4;23(1):72. doi: 10.1186/s13075-021-02453-7. PMID 33663558
- [Background] Borba AKOT, Arruda IKG, Marques APO, Leal MCC, Diniz ADS. Knowledge and attitude about diabetes self-care of older adults in primary health care. Cien Saude Colet. 2019 Jan;24(1):125-136. doi: 10.1590/1413-81232018241.35052016. English, Portuguese. PMID 30698247
- [Background] Nassar CM, Montero A, Magee MF. Inpatient Diabetes Education in the Real World: an Overview of Guidelines and Delivery Models. Curr Diab Rep. 2019 Sep 12;19(10):103. doi: 10.1007/s11892-019-1222-6. PMID 31515653
- [Background] Guarnaccia S, Quecchia C, Festa A, Magoni M, Moneda M, Gretter V, Scarcella C, Pluda A, Gasparotti C, Frassine M, Vitale L, D'Agata E, Limina RM, Donato F. Evaluation of a diagnostic therapeutic educational pathway for asthma management in youth. Pediatr Allergy Immunol. 2018 Mar;29(2):180-185. doi: 10.1111/pai.12839. Epub 2017 Dec 19. PMID 29168239
- See also: NATIONAL INSTITUTE OF HEALTH AND MEDICAL RESEARCH (INSERM). Sclérose en plaques (SEP) : Une recherche active pour améliorer la prise en charge des patients — https://www.inserm.fr/dossier/sclerose-en-plaques-sep/
- See also: PETER, Mireille and DE BRUYCKER, Christelle. L'éducation thérapeutique du patient dans la SEP: Place au patient. In: Le Courrier de la SEP, May 2015, No. 143. CHRU de Lille. — https://dumas.ccsd.cnrs.fr/dumas-01799522/document
- See also: BERTIN, Juliette and GENTY, Margot. Place de l'éducation thérapeutique dans la prise en charge de la sclérose en plaques. [online]. Paris Academy, University Paris VI Pierre and Marie Curie, academic year 2014-2015. — https://dumas.ccsd.cnrs.fr/dumas-01212307/document
- See also: PATHAK, Lokesh. Personalized Treatment for Multiple Sclerosis: The Role of Precision Medicine. Neurology Letters, 2023, vol. 2, no 1, p. 30-34. — https://www.neurologyletters.com/article_170305_9fb537f166dd3c37f265a9c50996bc2a.pdf